CLINICAL TRIAL: NCT00470704
Title: A Phase 2 Study of Lapatinib in Combination With Trastuzumab in Patients With HER2-Positive, Metastatic Breast Cancer
Brief Title: Lapatinib in Combination With Trastuzumab in Patients With HER2-Positive, Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nancy Lin, MD (Other)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Nancy Lin, MD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-213
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Results first posted 2022-03-15 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: HER2-positive breast cancer; Herceptin; trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Other): This cohort is made up of participants without prior trastuzumab for MBC. Adjuvant or neoadjuvant trastuzumab was allowed, if the interval from trastuzumab completion to recurrence exceeded 1 year.
  1000 mg daily Lapatinib
  2 mg/kg weekly or 6 mg/kg every 3 week dose of trastuzumab
  Interventions: Drug: Lapatinib; Drug: Herceptin
- Cohort 2 (Other): This cohort is made up of participants with one to two lines of chemotherapy for metastatic disease with at least one trastuzumab-containing regimen or patients who recurred within 12 months of adjuvant or neoadjuvant trastuzumab with up to one line of metastatic trastuzumab-based therapy
  1000 mg daily Lapatinib
  2 mg/kg weekly or 6 mg/kg every 3 week dose of trastuzumab
  Interventions: Drug: Lapatinib; Drug: Herceptin

INTERVENTIONS:
Drug: Lapatinib
  Other Names: Tykerb
Drug: Herceptin
  Other Names: trastuzumab

SUMMARY:
In this research study we are studying the effects of the combination of lapatinib plus Herceptin in subjects with breast cancer that has spread outside of the breast. We are also studying whether positron emission tomography (PET/CT) scans can predict which participants will benefit from the study treatment. Finally, we are studying genes and proteins in the tumor tissue that may lead to sensitivity or resistance to Herceptin, and to the combination of Herceptin plus lapatinib. Lapatinib is a compound that may stop cancer cells from growing. Other research studies suggest that lapatinib in combination with Herceptin may help to shrink or stabilize breast cancer.

DETAILED DESCRIPTION:
* Participants will be asked to undergo a biopsy of an area of the body where the cancer has spread.
* Participants will be given a study medication-dosing calendar for each treatment cycle. Each treatment cycle lasts four weeks during which time you will be taking lapatinib, once per day.
* Participants will receive Herceptin once every week or once every 3 weeks through a vein.
* During all treatment cycles a physical exam will be performed and questions about the participants general health will be asked. Blood tests including chemistry and hematology will be performed to measure additional effect of the study drug and disease status. Photographs may be taken of the tumor to assess the response of the tumor to treatment.
* CT scans will be repeated every 8 weeks to assess the effect of the study treatment on the cancer. Either a MUGA scan or echocardiogram will be performed 8 weeks and 16 weeks after the participant starts the study treatment.
* Participants will remain on this research study for as long as they are benefiting from the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer, with stage IV disease
* HER2-positive breast cancer, defined as 3+ staining by IHC or gene amplification by FISH
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension
* Willingness to undergo a research biopsy of recurrent or metastatic disease
* Prior chemotherapy treatment must be discontinued for at least 2 weeks prior to study entry.
* Completed radiation therapy at least 7 days prior to beginning protocol treatment
* Cohort 1: No prior chemotherapy for advanced breast cancer; no prior trastuzumab in the advanced breast cancer setting; nor prior treatment with lapatinib or other HER2-directed therapy other than trastuzumab
* Cohort 2: Up to two prior chemotherapy regimens for the treatment of advanced breast cancer; no prior treatment with lapatinib or other HER2-directed therapy except for trastuzumab
* 18 years of age or older
* Life expectancy of greater than 12 weeks
* ECOG Performance Status 0-2
* Normal organ and marrow function as outlined in protocol
* Cardiac ejection fraction, as assessed by either MUGA scan or echocardiogram greater than or equal to 50%
* Able to take oral medications

Exclusion Criteria:

* Patients may not be receiving any other investigational agents or concurrent chemotherapy or hormonal therapy for treatment of metastatic disease
* Active brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib or other agents used in this study
* Clinically significant malabsorption syndrome
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding women
* Concurrent use of the medications listed in the protocol because of possible interaction with lapatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-05-14 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2024-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - University fo Alabama at Birmingham, Birmingham, Alabama
  - University of Chicago, Chicago, Illinois
  - Dana-Farber at Faulkner Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin NU, Guo H, Yap JT, Mayer IA, Falkson CI, Hobday TJ, Dees EC, Richardson AL, Nanda R, Rimawi MF, Ryabin N, Najita JS, Barry WT, Arteaga CL, Wolff AC, Krop IE, Winer EP, Van den Abbeele AD. Phase II Study of Lapatinib in Combination With Trastuzumab in Patients With Human Epidermal Growth Factor Receptor 2-Positive Metastatic Breast Cancer: Clinical Outcomes and Predictive Value of Early [18F]Fluorodeoxyglucose Positron Emission Tomography Imaging (TBCRC 003). J Clin Oncol. 2015 Aug 20;33(24):2623-31. doi: 10.1200/JCO.2014.60.0353. Epub 2015 Jul 13. PMID 26169615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Registered between May 2007 and October 2010.
Groups:
- Cohort 1: This cohort is made up of participants without prior trastuzumab for MBC. Adjuvant or neoadjuvant trastuzumab was allowed, if the interval from trastuzumab completion to recurrence exceeded 1 year.
  1000 mg daily Lapatinib
  2 mg/kg weekly or 6 mg/kg every 3 week dose of trastuzumab
  Lapatinib: Oral dose taken daily
  Herceptin: Given intravenously once a week or once every 3 weeks
- Cohort 2: This cohort is made up of participants with one to two lines of chemotherapy for metastatic disease with at least one trastuzumab-containing regimen or patients who recurred within 12 months of adjuvant or neoadjuvant trastuzumab with up to one line of metastatic trastuzumab-based therapy
  1000 mg daily Lapatinib
  2 mg/kg weekly or 6 mg/kg every 3 week dose of trastuzumab
  Lapatinib: Oral dose taken daily
  Herceptin: Given intravenously once a week or once every 3 weeks
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 41 | 46
Safety Population | 41 | 45
Treated | 40 | 45
Completed | 0 | 0
Not Completed | 41 | 46
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Relapse/Progression | 37 | 42
Not completed — toxicity | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 41 | 45 | 86
Age, Continuous [Median (Full Range); unit: years] | 55 [32 to 77] | 50 [33 to 83] | 52 [32 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 86
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 35 | 43 | 78
  Unknown or Not Reported | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36 | 43 | 79
  Black and African American | 2 | 2 | 4
  Asian | 1 | 0 | 1
  Other | 2 | 0 | 2
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants]
  00 - Fully Active | 26 | 30 | 56
  01 - Restricted | 14 | 14 | 28
  02 - Ambulatory | 1 | 1 | 2
Stage at Initial Diagnosis [Count of Participants; unit: Participants] — Stage I: Cancer in the breast only, or tumor smaller than 2 cm in diameter with lymph node cancer cell groups of 0.2mm to 2mm in diameter.
  Stage II: Cancer has either spread to the lymph nodes or is 2cm - 5cm in diameter and human epidermal growth factor receptor 2 positive.
  Stage III: Cancer may spread to the skin or breast, or infected 4+ axillary lymph nodes or beyond the axillary lymph nodes or near the breastbone.
  Stage IV: Cancer has spread to other areas of the body, such as the brain, bones, lung and liver
  Participants
    Stage I | 4 | 5 | 9
    Stage II | 11 | 11 | 22
    Stage III | 10 | 18 | 28
    Stage IV | 16 | 9 | 25
    Unknown | 0 | 2 | 2
Hormone Receptor Status [Count of Participants; unit: Participants]
  Primary Tumor: Estrogen Receptor Positive and/or Progesterone Positive | 27 | 25 | 52
  Primary Tumor: Estrogen Receptor Negative and Progesterone Receptor Negative | 13 | 19 | 32
  Primary Tumor: Unknown or Not Done | 1 | 1 | 2
  Metastatic Lesion: Estrogen Receptor Positive and/or Progesterone Positive | 16 | 25 | 41
  Metastatic Lesion: Estrogen Receptor Negative and Progesterone Receptor Negative | 17 | 16 | 33
  Metastatic Lesion: Unknown or Not Done | 8 | 4 | 12
Human Epidermal Growth Factor Receptor 2 [Count of Participants; unit: Participants]
  Primary Tumor: Positive | 33 | 37 | 70
  Primary Tumor: Negative / Equivocal | 5 | 5 | 10
  Primary Tumor: Unknown / Not Done | 3 | 3 | 6
  Metastatic Lesion: Positive | 33 | 40 | 73
  Metastatic Lesion: Negative / Equivocal | 0 | 1 | 1
  Metastatic Lesion: Unknown / Not Done | 8 | 4 | 12
Disease-Free Interval [Count of Participants; unit: Participants]
  0 years (De Novo Metastatic Breast Cancer) | 16 | 9 | 25
  Greater than 2 years | 8 | 14 | 22
  Less than or equal to 2 years | 17 | 22 | 39
Median Number of Metastatic Disease Sites (Range) [Median (Full Range); unit: number of sites] | 3 [1 to 6] | 2 [1 to 5] | 3 [1 to 6]
Disease Sites [Count of Participants; unit: Participants]
  Central Nervous System | 1 | 5 | 6
  Lung | 20 | 12 | 32
  Pleural Effusion | 3 | 4 | 7
  Liver | 20 | 18 | 38
  Bone | 19 | 20 | 39
  Breast or Chest Wall | 22 | 24 | 46
  Lymph Nodes | 32 | 27 | 59
  Other | 6 | 5 | 11
Prior Therapy [Count of Participants; unit: Participants]
  Adjuvant or neoadjuvant hormonal therapy | 11 | 21 | 32
  Adjuvant or neoadjuvant chemotherapy | 19 | 27 | 46
  Anthracycline | 17 | 25 | 42
  Taxane | 14 | 24 | 38
  Trastuzumab | 8 | 21 | 29
Number of Lines of Chemotherapy for Metastasis or Recurrence [Count of Participants; unit: Participants]
  None | 39 | 7 | 46
  One | 1 | 20 | 21
  Two | 0 | 15 | 15
  Three | 1 | 3 | 4
Prior Chemotherapy for Metastasis or Recurrence [Count of Participants; unit: Participants]
  Trastuzumab | 1 | 38 | 39
  Trastuzumab-Emtansine | 1 | 0 | 1
  Pertuzumab | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The objective response rate is the percentage of participants achieving complete response (CR) or partial response (PR) as the best response recorded on treatment based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria.
  CR and PR must meet the following lesion criteria without having any new lesions as well:
  Target Lesion:
  (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Non-Target Lesion:
  (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  Non-CR/Non-Progressive Disease: Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. Must have PR in target lesion.
Time Frame: 8 weeks
Population: Given for all treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 40 | 45
percentage of participants | 50.0 [33.8 to 66.2] | 22.2 [11.3 to 37.3]

2. Secondary Outcome: Top 3 Most Common Treatment RelatedToxicities
Description: Assessed by -Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Top 3 treatment-related all-grade adverse events in terms of incidence.
  Treatment Related is discerned as follows:
  Yes: There is a plausible temporal relationship between the onset of the AE and administration of atezolizumab or bevacizumab, and the AE cannot be readily explained by the patient's clinical state, intercurrent illness, or concomitant therapies; and/or the AE follows a known pattern of response to atezolizumab or bevacizumab or with similar treatments; and/or the AE resolves upon discontinuation of the study drugs or dose reduction and, if applicable, reappears upon re-challenge.
  No: Evidence exists that the AE has an etiology other than the study drugs (e.g., pre existing medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the AE has no plausible temporal relationship to the study drugs administration.
Time Frame: Up to 93 months
Measure: Number; unit: toxicity events
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 40 | 45
toxicity events
  Diarrhea | 27 | 28
  Fatigue | 21 | 24
  Acne | 20 | 15

3. Secondary Outcome: Sites of First Progression
Description: Progression is defined by Response Evaluation Criteria In Solid Tumors Criteria 1.1 (RECIST) as follows:
  - >20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including baseline if it's the smallest). The sum must also demonstrate an increase of >5 mm.
  OR
  -Appearance of new lesions and/or unequivocal progression of non-target lesions. It must be representative of overall disease status change, not a single lesion increase. For patients with PD at the first on-treatment imaging assessment, patients will be allowed to remain on study until confirmation at the next assessment at investigator discretion if patient is benefiting from treatment.
Time Frame: Up to 93 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 41 | 46
Participants
  Central Nervous System (CNS) | 3 | 3
  Non-CNS | 31 | 39
  CNS and Non-CNS | 3 | 0
  NA | 4 | 4

4. Secondary Outcome: Clinical Benefit Rate
Description: Clinical Benefit Rate is the percentage of participants who achieve clinical benefit from the study treatment. Clinical benefit is defined as at least 24 weeks of confirmed Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
  SD or better is achieved if the following are true:
  Target Lesions:
  -At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Non-target Lesions:
  No progression. No appearance new lesions or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 93 months
Population: Given for all treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 40 | 25
percentage of participants | 57.5 [40.9 to 73] | 40.0 [25.7 to 55.7]

5. Secondary Outcome: 3-Year Overall Survival
Description: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive. 3-Year survival is calculated using Kaplan-Meier methods.
Time Frame: Up to 93 months
Population: Given for all treated patients
Measure: Number (95% Confidence Interval); unit: probability of survival
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 40 | 45
probability of survival | .62 [.47 to .81] | .39 [.26 to .57]

6. Secondary Outcome: Median Time to Progression
Description: Time to progression (TTP) is defined as the time from study entry to disease progression by RECIST. Subjects are considered to have progressed if they discontinue treatment due to clinical deterioration from breast cancer or die on-treatment of any cause. TTP is censored at the time of initiation of alternative therapy or time of last contact. The time to progression is calculated using a Kaplan-Meier emthods.
  Progression is defined by RECIST as:
  >20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including baseline if it's the smallest). The sum must also demonstrate an increase of >5 mm.
  OR Appearance of new lesions and/or unequivocal progression of non-target lesions. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 93 months
Population: Given for all treated patients
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 40 | 45
months | 7.4 [3.9 to 9.3] | 5.3 [3.7 to 6.7]

ADVERSE EVENTS:
Time Frame: Up to 93 months
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Groups:
- Cohort 1: This cohort is made up of participants without prior trastuzumab for MBC. Adjuvant or neoadjuvant trastuzumab was allowed, if the interval from trastuzumab completion to recurrence exceeded 1 year.
  1000 mg daily Lapatinib
  2 mg/kg weekly or 6 mg/kg every 3 week dose of trastuzumab
  Lapatinib
  Herceptin
- Cohort 2: This cohort is made up of participants with one to two lines of chemotherapy for metastatic disease with at least one trastuzumab-containing regimen or patients who recurred within 12 months of adjuvant or neoadjuvant trastuzumab with up to one line of metastatic trastuzumab-based therapy
  1000 mg daily Lapatinib
  2 mg/kg weekly or 6 mg/kg every 3 week dose of trastuzumab
  Lapatinib
  Herceptin
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 15/41 | 34/46
Serious Adverse Events (participants affected / at risk) | 2/41 | 7/46
Other Adverse Events (participants affected / at risk) | 40/41 | 44/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=41) | Cohort 2 (N=46)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 5
GI-other (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=41) | Cohort 2 (N=46)
Abdomen, pain (Gastrointestinal disorders) | 4 | 3
Alkaline phosphatase (Investigations) | 5 | 9
Alkalosis (Metabolism and nutrition disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Allergy-other (Immune system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2
ALT, SGPT (Investigations) | 12 | 11
Anorexia (Metabolism and nutrition disorders) | 8 | 7
Anxiety (Psychiatric disorders) | 8 | 6
Arachnoiditis/meningismus/radiculitis (Nervous system disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 4
AST, SGOT (Investigations) | 15 | 15
Ataxia (Nervous system disorders) | 3 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 9 | 8
Bicarbonate (Metabolism and nutrition disorders) | 0 | 4
Bilirubin (Investigations) | 2 | 3
Bone, pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Brachial plexopathy (Nervous system disorders) | 0 | 1
Breast, pain (Reproductive system and breast disorders) | 3 | 2
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 1 | 0
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Chest/thoracic pain NOS (General disorders) | 2 | 2
Cognitive disturbance (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 4
Constitutional, other (General disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4
C-P arrest, non-fatal, cause unknown (Cardiac disorders) | 1 | 0
Creatinine (Investigations) | 3 | 2
Depression (Psychiatric disorders) | 1 | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 28 | 30
Distention/bloating, abdominal (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 7 | 4
Dry eye syndrome (Eye disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 5 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Edema limb (General disorders) | 5 | 2
Edema trunk/genital (General disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 2
Extremity upper (function) (Musculoskeletal and connective tissue disorders) | 0 | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Extremity-lower (gait/walking) (General disorders) | 1 | 0
Fatigue (General disorders) | 23 | 30
Fever w/o neutropenia (General disorders) | 4 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 2
GI10 (Gastrointestinal disorders) | 1 | 0
gi111 (Gastrointestinal disorders) | 1 | 0
GI-other (Gastrointestinal disorders) | 1 | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1 | 5
Head/headache (Nervous system disorders) | 13 | 6
Hearing-other (Ear and labyrinth disorders) | 1 | 0
Hematologic-other (Blood and lymphatic system disorders) | 0 | 2
Hemoglobin (Blood and lymphatic system disorders) | 14 | 8
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Hemorrhage-other (Vascular disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 3 | 0
Hepatic-other (Hepatobiliary disorders) | 1 | 0
Hot flashes (Vascular disorders) | 5 | 6
Hyopthyroidism (Endocrine disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolemia (Investigations) | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 15
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 12 | 4
Hyperthyroidism, thyrotoxicosis (Endocrine disorders) | 2 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3
Hyponatremia (Metabolism and nutrition disorders) | 3 | 4
Hypotension (Vascular disorders) | 0 | 1
Infection Gr0-2 neut, lip/perioral (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, sinus (Infections and infestations) | 1 | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1 | 2
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 1 | 0
Infection w/ unk ANC bladder (Infections and infestations) | 1 | 0
Infection w/ unk ANC lung (Infections and infestations) | 1 | 1
Infection w/ unk ANC middle ear (Infections and infestations) | 1 | 0
Infection w/ unk ANC sinus (Infections and infestations) | 2 | 0
Infection w/ unk ANC ungual (nails) (Infections and infestations) | 1 | 0
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 2 | 1
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 0 | 1
Infection-other (Infections and infestations) | 4 | 2
Insomnia (Psychiatric disorders) | 8 | 3
Intra-op injury Other (Specify) (Injury, poisoning and procedural complications) | 1 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Keratitis (Eye disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0
Leukocytes (Investigations) | 1 | 4
Liver, pain (Hepatobiliary disorders) | 0 | 1
Lymph node, pain (Blood and lymphatic system disorders) | 1 | 0
Lymphatics-other (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Investigations) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Metabolic/Laboratory-other (Investigations) | 3 | 3
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1 | 1
Muco/stomatitis by exam, larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 6 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 0 | 3
Muscle, pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1 | 4
Nail changes (Skin and subcutaneous tissue disorders) | 9 | 3
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 11 | 17
Neck, pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Neurologic-other (Nervous system disorders) | 1 | 2
Neuropathy CN III pupil/eyelid/extraocul (Nervous system disorders) | 1 | 0
Neuropathy-motor (Nervous system disorders) | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 5 | 7
Neutrophils (Investigations) | 3 | 2
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Ocular-other (Eye disorders) | 4 | 3
Oral cavity, pain (Gastrointestinal disorders) | 1 | 1
Pain NOS (General disorders) | 0 | 1
Pain-other (General disorders) | 1 | 3
Palpitations (Cardiac disorders) | 0 | 1
Pelvic, pain (Reproductive system and breast disorders) | 1 | 1
Platelets (Investigations) | 0 | 2
Portal vein flow (Hepatobiliary disorders) | 0 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 | 6
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 | 7
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 21 | 16
Rectum, hemorrhage (Gastrointestinal disorders) | 1 | 0
Renal/GU-other (Renal and urinary disorders) | 2 | 0
Rigors/chills (General disorders) | 2 | 0
Sinus, pain (Nervous system disorders) | 1 | 0
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin, pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin-other (Skin and subcutaneous tissue disorders) | 5 | 1
Stomach, pain (Gastrointestinal disorders) | 2 | 2
Sweating (Skin and subcutaneous tissue disorders) | 1 | 1
Taste disturbance (Nervous system disorders) | 2 | 0
Teeth (Gastrointestinal disorders) | 1 | 0
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Vagina, hemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 1 | 2
Vasovagal episode (Nervous system disorders) | 0 | 1
Vision-blurred (Eye disorders) | 2 | 1
Vision-flashing lights/floaters (Eye disorders) | 0 | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 9 | 8
Weight gain (Investigations) | 1 | 1
Weight loss (Investigations) | 1 | 0
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes